CLINICAL TRIAL: NCT00390286
Title: Telemedicine's Utility for Augmenting Clinical Trials and Informed Consent TACTIC
Status: Withdrawn | Type: Observational
Why Stopped: no funding
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Brett Meyer, MD, University of California, San Diego
Other Study IDs: 051010
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Stroke
Keywords: Telemedicine
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a 6 year, Phase I, Clinical Research Protocol to study the feasibility of using a telemedicine system for performing research in a remote hospital system.

DETAILED DESCRIPTION:
The UCSD Telemedicine system is a digital video camera system, which can transfer video and audio images from a clinic or emergency room to a remote place where a physician can review images in real time (as they happen). The system uses site independent software to access the camera system from multiple locations. This research study will determine if it is feasible to obtain informed consent for various types of research trials (hypothetical, non-invasive, invasive trails) via telemedicine. Inpatient assessments on participants to complete clinical research case report forms by telemedicine will also by performed.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female, age 18 years or older
* Clinical neurological focal deficits consistent with stroke
* Time of onset 3-24 hours and with stable neurological deficit
* Signed Informed Consent

Exclusion Criteria:

* Deficits known to be due to non-stroke etiology
* Time of onset less than 3 hours
* Patients unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute stroke patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2019-12 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Number of trials participant is enrolled into | 5 years
  Counting how many patients are enrolled into OTHER clinical trials using a telemedicine technique

CONTACTS AND LOCATIONS:
Overall Officials: Brett C. Meyer, MD, Principal Investigator — UCSD Medical Center
Locations (1):
- UCSD Stroke Center, San Diego, California, United States

REFERENCES:
- [Background] Meyer BC, Lyden PD, Al-Khoury L, Cheng Y, Raman R, Fellman R, Beer J, Rao R, Zivin JA. Prospective reliability of the STRokE DOC wireless/site independent telemedicine system. Neurology. 2005 Mar 22;64(6):1058-60. doi: 10.1212/01.WNL.0000154601.26653.E7. PMID 15781827
- [Background] LaMonte MP, Bahouth MN, Hu P, Pathan MY, Yarbrough KL, Gunawardane R, Crarey P, Page W. Telemedicine for acute stroke: triumphs and pitfalls. Stroke. 2003 Mar;34(3):725-8. doi: 10.1161/01.STR.0000056945.36583.37. Epub 2003 Jan 30. PMID 12624298
- [Background] Levine SR, Gorman M. "Telestroke" : the application of telemedicine for stroke. Stroke. 1999 Feb;30(2):464-9. doi: 10.1161/01.str.30.2.464. PMID 9933289
- [Background] Audebert HJ, Kukla C, Clarmann von Claranau S, Kuhn J, Vatankhah B, Schenkel J, Ickenstein GW, Haberl RL, Horn M; TEMPiS Group. Telemedicine for safe and extended use of thrombolysis in stroke: the Telemedic Pilot Project for Integrative Stroke Care (TEMPiS) in Bavaria. Stroke. 2005 Feb;36(2):287-91. doi: 10.1161/01.STR.0000153015.57892.66. Epub 2004 Dec 29. PMID 15625294
- [Background] Wiborg A, Widder B; Telemedicine in Stroke in Swabia Project. Teleneurology to improve stroke care in rural areas: The Telemedicine in Stroke in Swabia (TESS) Project. Stroke. 2003 Dec;34(12):2951-6. doi: 10.1161/01.STR.0000099125.30731.97. Epub 2003 Nov 20. PMID 14631092
- [Background] Wang S, Gross H, Lee SB, Pardue C, Waller J, Nichols FT 3rd, Adams RJ, Hess DC. Remote evaluation of acute ischemic stroke in rural community hospitals in Georgia. Stroke. 2004 Jul;35(7):1763-8. doi: 10.1161/01.STR.0000131858.63829.6e. Epub 2004 May 27. PMID 15166386
- [Derived] Meyer BC, Raman R, Chacon MR, Jensen M, Werner JD. Reliability of site-independent telemedicine when assessed by telemedicine-naive stroke practitioners. J Stroke Cerebrovasc Dis. 2008 Jul-Aug;17(4):181-6. doi: 10.1016/j.jstrokecerebrovasdis.2008.01.008. PMID 18589337